CLINICAL TRIAL: NCT01784003
Title: Characterizing Ankle Function During Sloped Locomotion for Prosthesis Development
Status: Completed | Type: Observational
Sponsor: VA Eastern Colorado Health Care System (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: A7972W
Record Dates: First submitted 2013-01-25; First posted 2013-02-05 (Estimated); Last update posted 2020-09-10 (Actual); Status verified 2020-09

CONDITIONS: Traumatic Amputation of Lower Extremity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional

GROUPS / COHORTS (2):
- Non-amputee: People without an amputation will be recruited to participate in the study.
- Below the knee amputee: People with a unilateral transtibial amputation will be recruited to participate in the study.
  Interventions: Device: Powered ankle-foot prosthesis

INTERVENTIONS:
Device: Powered ankle-foot prosthesis
  Groups: Below the knee amputee

SUMMARY:
The proposed study aims to characterize biological ankle joint function during walking and running on slopes in order to further develop advanced powered ankle-foot prostheses. Ankle joint torque and angle data will be collected from non-amputees while walking and running at multiple speeds and slopes. This data will be used to develop control parameters for a powered ankle-foot prosthesis. Then, these parameters will be implemented and tested in a powered prosthesis worn by people with below the knee amputations.

ELIGIBILITY:
Inclusion Criteria:

Study 1:

- Between 18-60 years old.

Study 2 and 3:

* Between 18-60 years old.
* At least 1 year post-amputation
* no current problems with prosthesis or residual limb
* At least a K3 level of ambulation

Study 4:

- Between 18-45 years old

Study 5:

* Between 18-45 years old
* At least 1 year post-amputation
* no current problems with prosthesis or residual limb
* Experience running with a passive prosthesis
* At least a K4 level of ambulation

Exclusion Criteria:

Studies 1-5

* Cardiovascular, pulmonary, or neurological disease or disorder
* Musculoskeletal injury

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Study 1: Non-amputee Study 2: Unilateral transtibial amputee Study 3: Unilateral transtibial amputee Study 4: Non-amputee Study 5: Unilateral transtibial amputee
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2012-06; Primary Completion 2020-09 (Actual); Study Completion 2020-09 (Actual)

PRIMARY OUTCOMES:
Force-measuring treadmill and motion capture | approximately 2 months
Metabolic analysis system | approximately 2 months

CONTACTS AND LOCATIONS:
Locations (1):
- University of Colorado Boulder, Boulder, Colorado, United States

REFERENCES:
- [Result] Jeffers JR, Auyang AG, Grabowski AM. The correlation between metabolic and individual leg mechanical power during walking at different slopes and velocities. J Biomech. 2015 Aug 20;48(11):2919-24. doi: 10.1016/j.jbiomech.2015.04.023. Epub 2015 Apr 22. PMID 25959113
- [Result] Montgomery JR, Grabowski AM. The contributions of ankle, knee and hip joint work to individual leg work change during uphill and downhill walking over a range of speeds. R Soc Open Sci. 2018 Aug 29;5(8):180550. doi: 10.1098/rsos.180550. eCollection 2018 Aug. PMID 30225047
- [Result] Pickle NT, Grabowski AM, Jeffers JR, Silverman AK. The Functional Roles of Muscles, Passive Prostheses, and Powered Prostheses During Sloped Walking in People With a Transtibial Amputation. J Biomech Eng. 2017 Nov 1;139(11):1110051-11100511. doi: 10.1115/1.4037938. PMID 28975280
- [Result] Pickle NT, Grabowski AM, Auyang AG, Silverman AK. The functional roles of muscles during sloped walking. J Biomech. 2016 Oct 3;49(14):3244-3251. doi: 10.1016/j.jbiomech.2016.08.004. Epub 2016 Aug 6. PMID 27553849
- [Result] Montgomery JR, Grabowski AM. Use of a powered ankle-foot prosthesis reduces the metabolic cost of uphill walking and improves leg work symmetry in people with transtibial amputations. J R Soc Interface. 2018 Aug;15(145):20180442. doi: 10.1098/rsif.2018.0442. PMID 30158189
- [Result] Jeffers JR, Grabowski AM. Individual Leg and Joint Work during Sloped Walking for People with a Transtibial Amputation Using Passive and Powered Prostheses. Front. Robot. AI, 22 December 2017. https://doi.org/10.3389/frobt.2017.00072